# **Statistical Analysis Plan**

Study Code RP-6306-02

Edition Number

Version 1.0

Date

31 July 2024

# Phase 1 Study of the PKMYT1 Inhibitor RP-6306 in Combination with Gemcitabine for the Treatment of Advanced Solid Tumors (MAGNETIC Study)

Statistical Analysis Plan for RP-6306-02

Phase 1 Study of the PKMYT1 Inhibitor RP-6306 in Combination with Gemcitabine for the Treatment of Advanced Solid Tumors (MAGNETIC Study)



# TABLE OF CONTENTS

| LIST OF | ABBREVIATIONS | 6 |
|---------|---------------------------------------------------------------|----|
| 1. | INTRODUCTION | 9 |
| 2. | STUDY OBJECTIVES AND ENDPOINTS | 9 |
| 2.1. | Module 1 Objectives and Endpoints | 9 |
| 2.2. | Analysis Endpoints | 11 |
| 2.2.1. | Safety Endpoints | 11 |
| 2.2.2. | Efficacy Endpoints | 11 |
| 2.2.3. | Pharmacokinetics | 12 |
| 2.2.4. | Biomarker endpoints | 12 |
| 3. | INVESTIGATIONAL PLAN | 12 |
| 3.1. | Overall Study Design and Plan | 12 |
| 3.2. | Schedule of Assessments | 14 |
| 3.2.1. | Dose and Schedule Finding | 16 |
| 3.2.2. | Maximum Tolerated Dose | 20 |
| 3.3. | Sample Size Considerations | 22 |
| 4. | ANALYSIS POPULATIONS | 22 |
| 4.1. | DLT Evaluable Population. | 22 |
| 4.2. | Efficacy Population | 22 |
| 4.3. | Safety Population | 23 |
| 4.4. | Pharmacokinetic Population | 23 |
| 5. | DATA AND ANALYSIS CONSIDERATIONS | 23 |
| 5.1. | General Principles | 23 |
| 5.2. | Study Day and Analysis Visit | 24 |
| 5.2.1. | Analysis Visit | 24 |
| 5.3. | Handling of Missing Data | 24 |
| 5.3.1. | Missing/Partial Dates in Adverse Events | 24 |
| 5.3.2. | Missing/Partial Dates in Concomitant Medication | 25 |
| 5.3.3. | Missing/Partial Dates during Screening Visit | 26 |
| 5.3.4. | Missing/Partial Dates in Post-study Anticancer Therapy | 26 |
| 5.3.5. | Missing/Partial Last Dose Date | 27 |
| 5.3.6. | Relationship and Severity Imputation Rules for Adverse Events | 28 |
| 6. | DISPOSITION, DEVIATIONS AND PATIENT CHARACTERISTIC DATA | 28 |

| 6.1. | Protocol Deviations | 28 |
|---|---|---|
| 6.2. | Demographic and Baseline Characteristics | 29 |
| 6.3. | Genotype and Mutation Status at Enrollment | 29 |
| 6.4. | Disease Characteristics | 29 |
| 6.5. | Medical History | 30 |
| 6.6. | Prior and Concomitant Medications | 30 |
| 7. | SAFETY AND EXPOSURE DATA | 31 |
| 7.1. | Adverse Events | 31 |
| 7.2. | Treatment Exposure | 33 |
| 7.3. | Laboratory Evaluations | 34 |
| 7.4. | Vital Signs and Abnormalities | 35 |
| 7.5. | 12-lead ECG | 36 |
| 7.6. | Physical Examination and ECOG Performance Status | 37 |
| 8. | EFFICACY DATA | 37 |
| 8.1. | Derivation of Efficacy Endpoints | 37 |
| 8.1.1. | Best Percentage Change in Tumor Size | 37 |
| 8.1.2. | Objective Response Rate (ORR) | 38 |
| 8.1.3. | Best Overall Response Rate | 38 |
| 8.1.4. | Clinical Benefit Rate (CBR) | 38 |
| 8.1.5. | Tumor marker response | 38 |
| 8.1.6. | Duration of Response (DOR) | 38 |
| 8.1.7. | Categorization of Best Tumor Response | 39 |
| 8.1.8. | Change in Tumor Size. | 39 |
| 8.1.9. | Progression Free Survival (PFS) | 40 |
| 8.2. | Efficacy Analysis Methods | 41 |
| 9. | PHARMACOKINETIC (PK) PARAMETERS DATA | 42 |
| 9.1. | Population PK/PD Modelling | 44 |
| 10. | BIOMARKER DATA | 44 |
| 11. | INTERIM ANALYSIS | 44 |
| 12. | REFERENCES | 45 |
| APPEND | DIX 1. DEFINITION OF DOSE LIMITING TOXICITY (DLT) | 46 |
| APPEND | OIX 2. GYNECOLOGICAL CANCER INTERGROUP DEFINITIONS FOR RESPONSE AND PROGRESSION IN PATIENTS WITH OVARIAN CANCER | 47 |

| Statist | ical A | nalysis | Plan |
|---------|--------|---------|-------|
| Study | Code | RP-630 | 06-02 |

| APPENDIX 3. | RESPONSE EVALUATION CRITERIA IN SOLID TUMORS, | |
|-------------|-----------------------------------------------|----|
| VFF | SION 1.1 | 40 |

# LIST OF ABBREVIATIONS

| Abbreviation or special term | Explanation |
|---|---|
| AE | Adverse Event |
| ADaM | Analysis Data Model |
| ALT | Alanine Aminotransferase |
| ALP | Alkaline Phosphatase |
| ANC | Absolute Neutrophil Count |
| AST | Aspartate Aminotransferase |
| AUC | Area Under the Curve |
| AUC0-8 | Area under the plasma concentration-time curve from time 0 to 8 hours post dose |
| AUC0-12 | Area under the plasma concentration-time curve from time 0 to 12 hours post dose |
| AUC0-inf | Area under the plasma concentration-time curve from time 0 to infinite time |
| AUC0-last | Area under the plasma concentration-time curve from time 0 to t ("t" being the longest time interval evaluable in all periods) |
| AUCss | Area under the plasma concentration-time curve at steady-state |
| BID | Twice daily |
| BOIN | Bayesian Optimal Interval |
| BP | Blood Pressure |
| BUN | Blood Urea Nitrogen |
| CBR | Clinical Benefit Rate |
| CCNE1 | Cyclin E1 |
| CDISC | Clinical Data Interchange Standards Consortium |
| CDK | Cyclin-dependent kinase |
| CDK1 | Cyclin-dependent kinase 1 |
| CDK2 | Cyclin-dependent kinase 2 |
| CI | Confidence Interval |
| C <sub>max</sub> | Maximum observed plasma Concentration |
| Cmin | Minimum observed plasma concentration |
| CR | Complete Response |
| CRF | Case Report Form |
| CSR | Clinical Study Report |
| CT | Computed Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| ctDNA | Circulating Tumor DNA |
| DBP | Diastolic Blood Pressure |

| Abbreviation or special term | Explanation |
|---|---|
| DCO | Data Cut off |
| DLT | Dose Limiting Toxicity |
| DNA | Deoxyribonucleic Acid |
| DOR | Duration of Response |
| ECG | Electrocardiogram |
| ECOG | Eastern Cooperative Oncology Group |
| eCRF | Electronic Case Report Form |
| ЕОТ | End-of-Treatment |
| FBXW7 | F-box and WD repeat domain containing 7 |
| FDA | Food and Drug Administration |
| FISH | Fluorescent in situ hybridization |
| GCP | Good Clinical Practice |
| G-CSF | Granulocyte Colony Stimulating Factor |
| GI | Gastrointestinal |
| ICF | Informed Consent Form |
| ICH | International Conference on Harmonization |
| IHC | Immunohistochemistry |
| LTFU | Lost to Follow-up |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Imaging |
| MTD | Maximal Tolerated Dose |
| NCA | Non-compartmental Analysis |
| NCI | National Cancer Institute |
| NE | Not Evaluable |
| NGS | Next-Generation Sequencing |
| ORR | Objective Response Rate |
| PD | Progressive Disease |
| PE | Physical Exam |
| PET | Positron Emission Tomography |
| PFS | Progression Free Survival |
| PK | Pharmacokinetics |
| PKMYT1 | Membrane-associated tyrosine- and threonine-specific Cdc2-inhibitory kinase |
| PODS | Precision Oncology Decision Support |
| PPP2R1A | Protein phosphatase 2 scaffold subunit A |
| PR | Partial Response |

| Abbreviation or special term | Explanation |
|---|---|
| PSA | Prostate-Specific Antigen |
| PT | Preferred Term |
| QD | Once daily |
| QT | ECG interval measured from the onset of the QRS complex to the end of the T wave |
| QTc | QT interval corrected for heart rate |
| QTcB | Bazett formula for corrected QT interval |
| QTcF | Fridericia formula for corrected QT interval |
| RBC | Red Blood Cells |
| RECIST | Response Evaluation Criteria in Solid Tumors |
| RP2D | Recommended Phase 2 Dose |
| SAE | Serious Adverse Event |
| SAP | Statistical Analysis Plan |
| SD | Stable Disease |
| SDTM | Study Data Tabulation Model |
| SOC | System Organ Class |
| SRC | Safety Review Committee |
| TEAE | Treatment Emergent Adverse Event |
| t½ | Terminal Elimination Half-Life |
| TL | Target Lesions |
| T <sub>max</sub> | Time to Maximum observed plasma concentration |
| ULN | Upper Limit of Normal |
| WBC | White Blood Cells |
| WHO | World Health Organization |

#### 1. INTRODUCTION

This statistical analysis plan (SAP) prospectively describes the planned analyses for the study Protocol RP-6306-02 "Phase 1 Study of the PKMYT1 Inhibitor RP-6306 in Combination with Gemcitabine for the Treatment of Advanced Solid Tumors (MAGNETIC Study)" Version 4.0, which was issued on 24 July 2023.

Due to closure of enrollment for Module 1c and 1d, this SAP will only cover the analyses for Module 1a and 1b.

The SAP is in full conformity with the most current version of Good Clinical Practices (GCP), the FDA and ICH Guidelines forclinical trials. It contains definitions of analysis populations, derived variables, and statistical methods for the analysis of efficacy and safety. In addition, the datasets generated for this study will be compliant with the latest version of the CDISC standards for the SDTM and ADaM datasets.

This SAP mainly covers the primary and secondary objectives of the study. Analyses for some of the exploratory objectives will be addressed outside the SAP, where additional analysis plans may be developed to address these objectives. In addition, population pharmacokinetics (PK) and PK/pharmacodynamic modelling will be addressed outside of the SAP.

The purpose of this SAP is to ensure the credibility of the study findings by pre-specifying the statistical approaches to the analysis of study data prior to database lock. This SAP will be finalized and approved prior to the clinical database lock.

#### 2. STUDY OBJECTIVES AND ENDPOINTS

2.1. Module 1 Objectives and Endpoints

| <b>Primary Objectives</b> | Primary Endpoints |
|---|---|
| To assess the safety and tolerability of RP-6306 in combination with gemcitabine in patients with eligible, advanced solid tumors | Incidence and severity of treatment-emergent adverse events (TEAEs), laboratory assessments, vital signs, electrocardiograms (ECGs), and use of concomitant medications |
| To define the maximum tolerated dose (MTD) and recommended Phase 2 Dose (RP2D) and schedule of RP-6306 in combination with gemcitabine | Dose-limiting toxicities (DLTs) |



# 2.2. Analysis Endpoints

The objective table provides information on the study objectives and analysis endpoints, split by primary, secondary and exploratory. The following section summarizes the primary, secondary, and exploratory analysis endpoints split by type of endpoints (safety, efficacy, PK, and biomarker).

#### 2.2.1. Safety Endpoints

- DLTs
- Incidence of TEAEs, treatment related TEAEs, TEAEs leading to death, serious adverse events (SAEs), treatment related SAEs, TEAEs leading to study drug discontinuation, TEAEs leading to dose modifications (interruptions or reductions)
- Changes in clinical laboratory parameters (hematology, chemistry, urinalysis), CTCAE graded laboratory toxicities, vital signs, Eastern Cooperative Oncology Group (ECOG) performance status, ECG parameters including QTc, physical exams (PEs) and usage of concomitant medications

#### 2.2.2. Efficacy Endpoints

- **Best percentage change in tumor size**: defined as the largest decrease or smallest increase (in the absence of a decrease) in the sum of diameters of the target lesions (TLs) prior to progression or last evaluable assessment in the absence of progression. More details can be found in Section 8.1.1.
- Objective response rate (ORR): defined as the proportion of patients with confirmed best overall response of complete response (CR) or partial response (PR) (i.e., 2 subsequent responses of either CR or PR at least 4 weeks apart) according to RECIST v1.1. More details can be found in Section 8.1.2.
- **Best overall response rate**: defined as the proportion of patients with **confirmed or unconfirmed** response of CR or PR based on best overall response by investigators across all visits. Unconfirmed CR or PR will be defined as those patients with CR or PR only reported once in overall tumor assessment form by the Investigators according to RECIST 1.1.
- Clinical benefit rate (CBR): defined as the proportion of patients with a best overall response of CR or PR according to RECIST v1.1 based on Investigator's assessment, or ovarian patients with tumor marker response (GCIG for CA-125), or duration on treatment of at least 16 weeks without evidence of progression.
- Tumor marker response (only for ovarian patients with abnormal baseline CA-125): defined as having ≥ 50% reduction from baseline in CA-125 and confirmed in next assessment based on GCIG criteria.
- Duration of response (DOR, applicable only to patients with confirmed CR or PR): defined as the time interval between the date of the earliest qualifying response (CR or PR) and the date of disease progression or death (if death occurred within 12 weeks after last adequate tumor assessment), whichever occurs earlier.

- For patients who are alive without disease progression following response, DOR will be censored on the date of last evaluable tumor assessment or last follow-up for disease progression.
- For patient who dies in the absence of progression, and the death is >12 weeks after the
  last evaluable tumor assessment, will be censored for DOR at the date of their last
  evaluable tumor assessment.
- **Progression-free survival (PFS)**: defined as the time from the first day of study treatment administration (Day 1) to disease progression as defined by RECIST v1.1 or death from any cause.
  - Patients who are alive and free from disease progression will be censored at the date of their last tumor assessment.
  - Any patient who dies in the absence of progression, and the death is >12 weeks after the
    last evaluable tumor assessment, will be censored for PFS at the date of their last
    evaluable tumor assessment.

Detailed derivation of the endpoints can be found in Section 37.



#### 3. INVESTIGATIONAL PLAN

# 3.1. Overall Study Design and Plan

This is a multicenter, open-label, Phase 1 study to evaluate the safety and preliminary efficacy of RP-6306, a first-in-class PKMYT1 inhibitor, given on a continuous or intermittent schedule in

combination with gemcitabine for the treatment of patients with relapsed or refractory, advanced solid tumors. The study will follow a Bayesian optimal interval (BOIN) drug combination design to identify the MTD (dose level and dosing schedule for Module 1a, Module 1b, Module 1c, and/or Module 1d) of RP-6306 and gemcitabine. Backfill cohorts with specific molecular alterations or cancer types will be enrolled to further evaluate the PK, pharmacodynamic and mechanism of action of biomarkers, safety and tolerability, and preliminary efficacy of the combination, as agreed upon by the Investigators and Safety Review Committee (SRC). The totality of safety, PK, pharmacodynamic, and preliminary efficacy data from each module will be used to establish a preferred RP2D and schedule (Figure 1). Eligible patients must have a tumor harboring a CCNE1 amplification or deleterious mutation in FBXW7 or PPP2R1A or other genetic alterations with mechanistic rationale agreed upon by the Sponsor and the Investigator. These genomic alterations are hypothesized to be synthetic lethal with RP-6306 and in preclinical mouse models were shown to be markedly sensitive to the combination of RP-6306 and gemcitabine.

The study will follow a Bayesian optimal interval (BOIN) drug combination design to identify the MTD (dose level and dosing schedule for Module 1a, Module 1b, Module 1c, and/or Module 1d) of RP-6306 and gemcitabine. Backfill cohorts with specific molecular alterations or cancer types will be enrolled to further evaluate the PK, pharmacodynamic and mechanism of action of biomarkers, safety and tolerability, and preliminary efficacy of the combination, as agreed upon by the Investigators and Safety Review Committee (SRC). The totality of safety, PK, pharmacodynamic, and preliminary efficacy data from each module will be used to establish a preferred RP2D and schedule.

Figure 1: Module 1 Study Schema



CCNE1=Cyclin E1; DLT=dose-limiting toxicity; FBXW7=F-box and WD repeat domain containing 7; PPP2R1A=protein phosphatase 2 scaffold subunit A; QD=once daily; RP2D=recommended Phase 2 Dose.

Note: Additional schedules may be tested based on safety, tolerability, and drug exposure data generated in all modules.

#### 3.2. Schedule of Assessments

The study will consist of a Screening Period (Day -28 to Day -1, to determine eligibility), a Treatment Period (21-day cycles), an End-of-Treatment (EOT) Period (occurring within 7 days after the last dose of study treatment), and a Safety Follow-up Period (occurring 30 days  $\pm$  2 weeks after the last dose of study

treatment for all patients not cleared at the EOT Visit, including patients with ongoing Grade ≥2 drug-related toxicities at the EOT Visit) (Figure 2).

Figure 2: Study Conduct



C1D1=Cycle1 Day 1; ctDNA=circulating tumor deoxyribonucleic acid; ECG=electrocardiogram; EOT=End-of-Treatment; FU=Follow-up; PD=progressive disease; PK=pharmacokinetic; RP2D=recommended Phase 2 dose

The start of the study is defined as the date when the first patient in the whole study signs an informed consent form (ICF).

The end of the study is defined as the date of the last visit (including all follow-up visits) of the last patient in the whole study.

See protocol for full details on the schedule of assessments.

The key procedures required in this study include:

- Tumor assessments (based on CT, PET, and/or MRI scan) according to RECIST v1.1 or as clinically indicated
- PK samples throughout the study
- Baseline, on-treatment, and EOT blood samples
- Reporting all AEs occurring from the administration of the first dose of RP-6306 and/or gemcitabine
- Paired-tumor biopsies

#### ECG

A cycle of treatment is 3 weeks (21 calendar days). Multiple procedures may be scheduled at the same timepoint relative to RP-6306 and gemcitabine dosing.

#### 3.2.1. Dose and Schedule Finding

This study aims to identify the RP2D and preferred dosing schedule of RP-6306 in combination with gemcitabine. RP-6306 will be given on a continuous schedule (Modules 1a and intermittent schedule (Modules 1b as a outlined below. Once triggered, Module 1b, and proceed concurrently with Module 1a, and escalation and de-escalation will proceed independently as guided by the BOIN drug combination criteria. Patients will be enrolled into Modules 1a, 1b, and d based on available slot openings at the time of signing the ICF and allocated to a cohort by the Medical Monitor with guidance from the SRC.

#### Module 1a

The study will start at Dose Level 1A with 1 patient receiving 40 mg QD, oral RP-6306 in combination with 800 mg/m² IV gemcitabine given over 30 minutes on Days 1 and 8 of each 21-day cycle. Upon clearing Dose Level 1A, Dose Level 2A will be initiated at 120 mg QD oral RP-6306 in combination with 800 mg/m² IV gemcitabine given over 30 minutes on Days 1 and 8 of each 21-day cycle. These dose levels of RP-6306 were chosen based on the observed tolerability of RP-6306 monotherapy in the MYTHIC study.

Dose escalation will proceed to the next higher dose level (Dose Level 3A) following BOIN criteria and dose escalation and de-escalation rules as follows:

- Dose escalation will progress with increases of up to 100% RP-6306 until a DLT is observed (Level R in Figure 3 and Table 1 presented below). Dose decisions will depend on 2 or more evaluable patients completing the first 21-day treatment cycle.
- After Level R, RP-6306 will be de-escalated per BOIN drug combination criteria. For de-escalation at Level R, the next dose level of RP-6306 will be ≥25% lower than the current dose (rounded down based on capsule strength) or de-escalated down to the highest previously tolerated dose based on review of the toxicity patterns by the SRC. Gemcitabine can be de-escalated up to 25%. Only one drug in the combination will be de-escalated at any time. In addition to decreasing the daily dose level of RP6306, de-escalation can involve a reduced frequency of dosing (eg, 5 days instead of planned 7 days or 2 days of RP-6306 rather than 3 days at the same dose level).
- After Level R, any dose escalation of RP-6306 or gemcitabine will follow the BOIN drug combination criteria as guided by the SRC. RP-6306 can continue with increases of 20% to 50% (R+1#), and dose escalation of gemcitabine can continue to a maximum of 1000 mg/m². Only 1 drug in the combination will be escalated at any time.

#### Module 1b

Module 1b will be initiated after the first DLT is observed in Module 1a. In Module 1b, an intermittent dosing schedule of RP-6306 given 3 consecutive days on / 4 consecutive days off will be tested in combination with gemcitabine if confirmed safe by the SRC. When Module 1b is initiated, the starting

dose of RP-6306 and gemcitabine will be the same as the highest total daily dose evaluated in Module 1a and will be given to a cohort of  $N\geq 2$ .





BOIN=Bayesian optimal interval; DLT=dose-limiting toxicity; MTD=maximum tolerated dose; QD=once daily.

| Table 1: | Dose Finding Phase |
|----------|--------------------|
|----------|--------------------|

| Table 1. | Dose II | nuing I na | | |
|---|---|---|---|---|
| | Module 1a <sup>a</sup> :<br>Contin | TO A CONTROL OF THE PARTY OF TH | Module 1b <sup>a</sup> : RP-6306 3 Consecutive Days On / 4 Consecutive Days Off | |
| Dose<br>Level | Total Daily RP-6306 Dose or % of Previous Dose | Gem<br>Dose<br>and<br>Schedule | Total Daily RP-6306 Dose or % of Previous Dose | Gem<br>Dose<br>and<br>Schedule |
| 1D | 40 mg | 600<br>mg/m <sup>2</sup><br>Days 1<br>and 8 | 40 mg | 600<br>mg/m <sup>2</sup><br>Days 1<br>and 8 |
| 1A <sup>b</sup><br>Starting<br>Dose<br>Level | 40 mg | 800<br>mg/m <sup>2</sup><br>Days 1<br>and 8 | Ξ | |
| 2A <sup>b</sup> | Up to 100%<br>increase<br>until Level<br>R | 800<br>mg/m <sup>2</sup><br>Days 1<br>and 8 | Ξ | = |
| | | | | I |

| R<br>(DLT) | Expand<br>cohort or<br>de-escalate<br>per BOIN<br>drug<br>combination<br>criteria | Same as<br>current<br>dose<br>level | | ı |
|---|---|---|---|---|
| R+1° | 20%-50%<br>increase or<br>25%-100%<br>decrease per<br>BOIN drug<br>combination<br>criteria | Up to<br>1000<br>mg/m <sup>2</sup><br>Days 1<br>and 8 | Same dose<br>as<br>continuous<br>schedule for<br>3 days only | Up to<br>1000<br>mg/m <sup>2</sup><br>Days 1<br>and 8 |
| R+N <sup>c</sup> | 20%-50%<br>increase or<br>25%-100%<br>decrease per<br>BOIN drug<br>combination<br>criteria | Up to<br>1000<br>mg/m <sup>2</sup><br>Days 1<br>and 8 | Per BOIN<br>drug<br>combination<br>criteria | Up to<br>1000<br>mg/m <sup>2</sup><br>Days 1<br>and 8 |

Gem=gemcitabine, BOIN=Bayesian optimal interval, DLT=dose-limiting toxicity, MTD=maximum tolerated dose.

If Dose Level 1A is not tolerated in Module 1a, Dose Level 1D will be explored. At Dose Level 1D, RP-6306 will be given at 40 mg daily on a continuous schedule and gemcitabine will be administered as an IV infusion at 600 mg/m² over 30 minutes on Days 1 and 8 of each 21-day cycle. If Dose Level 1D is tolerated and deemed safe by the SRC, gemcitabine dose will be maintained at 600 mg/m² given on Days 1 and 8 of each cycle and escalation of RP-6306 will proceed in increments of 25% to 50% in a continuous schedule. In addition, if Dose Level 1A is not tolerated using a continuous schedule, that same starting dose of RP-6306 (40 mg) and gemcitabine (800 mg/m²) will be tested on a 3 consecutive days on / 4 consecutive days off dosing schedule.



R: Dose level at which pharmacologic activity observed

N: Any dose level after R+1

<sup>&</sup>lt;sup>a</sup> Modules 1a, 1b, 1c, and 1d may progress independently.

<sup>&</sup>lt;sup>b</sup> Dose Levels 1A or 2A may be already Level R if early treatment-related toxicity is observed.

<sup>&</sup>lt;sup>c</sup> The order of escalation (RP-6306 or gemcitabine) will be guided by BOIN drug combination criteria and agreed upon by the SRC.

#### 3.2.2. Maximum Tolerated Dose

The BOIN drug combination design will be employed to find the MTD of continuous RP6306 (Module 1a, or intermittent RP-6306 (Module 1b, or

The BOIN design uses the following rules, optimized to minimize the probability of incorrect dose assignment, to guide dose escalation/de-escalation:

- If the observed DLT rate at the current dose is ≤0.197 (<20%), escalate the dose to one of the 2 next higher dose levels (ie, 1 level increase of RP-6306 or 1 level increase of gemcitabine).
- If the observed DLT rate at the current dose is ≥0.298 (≥30%), de-escalate the dose to one of the 2 next lower dose levels (ie, 1 level decrease of RP-6306 or 1 level decrease of gemcitabine).
- · Otherwise, stay at the current dose.

Table 2: Dose Escalation/De-Escalation Rules for the BOIN Design

| | Number of Evaluable Patients at Current Dose Level | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Action | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12 |
| ↑ if number of<br>DLT ≤ | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1. | 1 | 2 | 2 |
| Stay current<br>dose if<br>number of<br>DLT = | NA | NA | NA | 1 | 1. | NA | 2 | 2 | 2 | 2 | 3 | 3 |
| ↓ if number<br>of DLT ≥ | 1. | Ī | 1 | 2 | 2 | 2 | 3 | 3 | 3 | 3 | 4 | 4 |
| Elim if<br>number of<br>DLT≥ | NA | NA | 3 | 3 | 3 | 4 | 4 | 4 | 5 | 5 | 6 | 6 |

BOIN = Bayesian optimal interval; \( \gamma = \text{increase}, \( \psi = \text{decrease}, \text{DLT} = \text{dose-limiting toxicity}, \text{Elim=eliminate}, \text{NA} = \text{not applicable}, \\ \text{dose cannot be eliminated until at least 3 patients have been treated} \)

Note: Number of DLT is the number of patients with at least 1 DLT. When none of the actions (ie, escalate, de-escalate or eliminate) is triggered, stay at the current dose for treating the next cohort of patients.

Dose finding starts at Dose Level 1A. The steps to implement the BOIN design are described as follows:

- 1. Patients in the first cohort are treated at Dose Level 1A.
- 2. To assign a dose to the next cohort of patients, conduct dose escalation/de-escalation according to the rule displayed in the Dose Escalation/De-Escalation Rules table (Table 2). More details are provided in the study protocol.

After the study is completed, results from all DLT-evaluable patients including the relevant backfill cohorts will be included to assess the MTD. The dose for which the isotonic estimate of the toxicity rate is closest to and no higher than 25% will be selected as the MTD (<u>Liu and Yuan, 2015</u>). This computation can be implemented by the shiny app "BOIN" available at http://www.trialdesign.org. The RP2D for RP-6306 and gemcitabine will be based on discussion between the Investigators and the Sponsor and will be either the established MTD or a dose lower than MTD based on the totality of the safety, PK, pharmacodynamics, and preliminary efficacy.

# 3.3. Sample Size Considerations

The approximate sample size planned for this study is 150. The sample size per module for the Dose Finding Phase is 36 evaluable patients in Modules 1a and 1b and 21 evaluable patients in Modules 1c and 1d (114 total evaluable patients). To allow 10% non-evaluable rate, the total sample size for the Dose Finding Phase would be 126. Approximately an additional 24 patients will be planned for backfill cohorts.

The population used for determination of DLTs will consist of patients who have met the minimum safety evaluation requirements of the study, and/or who have experienced a DLT at any time during the first treatment cycle. Minimum safety requirements will be met if, during Cycle 1 of treatment the patient receives at least 75% of planned total doses of RP-6306 for the evaluated schedule, 100% of planned doses of gemcitabine, completes all required safety evaluations per Schedule of Assessments, and are observed at least until the end of the first treatment cycle. Depending on the toxicity profile of the combination and the number of dose levels required to establish the MTD/RP2D, the actual study sample size may vary.

Note that the study was ended earlier and module 1c and 1d was not executed.

#### 4. ANALYSIS POPULATIONS

# 4.1. DLT Evaluable Population

**DLT Evaluable Population** will consist of patients who have met the minimum safety evaluation requirements of the study and/or who experience a DLT at any time during the initial 21 days of the study. Minimum safety requirements will be met if, during Cycle 1 of treatment, the patient receives at least 75% of planned total doses of RP-6306 for the evaluated schedule, 100% of planned doses of gemcitabine, completes all required safety evaluations per the Schedule of Assessments in the protocol, and is observed at least until Day 21 since the first dose of study treatment. This population will be applied to dose escalation decisions in both modules 1a and 1b.

# 4.2. Efficacy Population

#### The Efficacy Population will be defined as below:

All patients who received at least 1 dose of RP-6306 and **evaluable for RECIST response** or evaluable for tumor marker response (GCIG for CA-125), or without post-baseline tumor assessment but discontinued the treatment due to clinical progression or death prior to any post-baseline tumor assessment, and without major eligibility deviation.

#### **Modified Efficacy Population** will be defined as below:

All patients who received at least 1 dose of RP-6306 and **evaluable for RECIST response** or evaluable for tumor marker response (GCIG for CA-125), and without major eligibility deviation.

For both efficacy populations, **evaluable for RECIST response** means patients are required to have measurable disease at baseline and at least 1 post-baseline tumor assessment. For patients with ovarian cancer without measurable disease but with elevated baseline CA-125 levels (>70 kU/L) and two post-baseline CA-125 that are done 3 weeks apart will be considered as CA-125 response evaluable.

The modified efficacy population was added for exploratory purpose.

# 4.3. Safety Population

The **Safety Population**, used for the assessment of overall safety and tolerability, will consist of all patients who receive at least one dose of study treatment. Patients will be assessed for safety based on the dose level in which they are enrolled.



#### 5. DATA AND ANALYSIS CONSIDERATIONS

# 5.1. General Principles

All demography and safety data will be presented by the safety population, except for the DLT reporting which will be based on the DLT evaluable population. Assessment of anti-tumor activity will be based on the Efficacy Population and PK data will be presented by the PK Population.

Most of the analyses will be descriptive in nature. Unless stated otherwise, continuous variables will be summarized using descriptive statistics (number of patients, mean, standard deviation, median, lower and upper quartile, minimum and maximum values) and the number and percentage of patients will be used for categorical variables. In general, missing data will be considered as missing and will not be imputed. Unless stated otherwise, percentages will be calculated out of the number of patients in the relevant analysis population.

Baseline will be the last assessment of the variable under consideration prior to first dose of RP-6306.

Unless stated otherwise, safety and efficacy data will be presented by assigned dose/schedule.

After determination of RP2D dose(s), safety and efficacy data may also be summarized by grouping dose levels based on RP2D and clinical relevance.

All DLT rates will be summarized by the assigned initial dose levels.

Summary statistics will be presented to the following degree of precision unless otherwise specified:

| | Degree of Precision |
|---|---|
| Mean, Geometric mean, Median, Quartiles,<br>Confidence limit boundaries | One more decimal digit than the raw data. |
| Standard deviation, Standard error | Two more than the raw data, with maximum of 4 digits |
| Minimum, Maximum | The same decimal digit as the raw data. |
| Percentage | One decimal place. A percentage of 100% will be reported as 100%. Percentages of zero will be reported as 0. |

# 5.2. Study Day and Analysis Visit

Study Day will be calculated from the reference start date (defined as the date of first dose of study drug), and will be used to show start/stop day of assessments/events:

Study Day = (date of assessments/events - reference start date) if event/assessment is prior to the reference start;

Study Day = (date of assessments/events - reference start date + 1) if event/assessment is on or after the reference start.

There is no Study Day 0.

#### 5.2.1. Analysis Visit

Baseline value will be the latest non-missing result obtained on or before the first dose of study treatment. The nominal visits will be used as analysis visits for the purpose of summarizing data over scheduled visit. If visits are clearly defined, no windowing algorithm will be used. If the cycle data are not clearly identifiable, study day with a window will be used to define the visits.

All recorded data will be included in the listings.

# 5.3. Handling of Missing Data

There will be no imputation of incomplete or missing data other than the dates mentioned below. No imputation will be performed for missing data elements for by-patient listings. However, the imputation will be implemented for summary tabulations, when applicable.

#### 5.3.1. Missing/Partial Dates in Adverse Events

#### **Missing Data Imputation for Adverse Event Start Dates**

If the stop date is non-missing and the imputed start date is after the stop date, the stop date will be used as the start date.

- (1) Missing day only
- If the month and year are the same as the month and year of the first dose date, the first dose date will be used.
- If the month and year are before the month and year of the first dose date, the last day of the month will be assigned to the missing day.
- If the month and year are after the month and year of the first dose date, the first day of the month will be assigned to the missing day.
- (2) Missing day and month
  - If the year is the same as the year of the first dose date, the first dose date will be used.
- If the year is prior to the year of the first dose date, December 31 will be assigned to the missing fields.
- If the year is after the year of the first dose date, January 1st will be assigned to the missing fields.

- (3) Missing day, month, and year (or only year)
  - The first dose date will be used.

#### Missing Data Imputation for Missing Adverse Event Stop Date

If the start date is non-missing and the imputed stop date is before the start date, the start date will be used. If the death date is available and the imputed stop date is after the death date, the death date will be used.

- (1) Missing day only
  - The last day of the month will be assigned as the missing day.
- (2) Missing day and month
  - December 31 will be assigned to the missing fields.
- (3) Missing day, month, and year (or only year)
  - The event will be regarded as ongoing.

#### **5.3.2.** Missing/Partial Dates in Concomitant Medication

#### **Missing Data Imputation for Concomitant Medication Start Dates**

If the stop date is non-missing and the imputed start date is after the stop date, the stop date will be used as the start date.

- (1). Missing day only
  - If the month and year are the same as the month and year of the first dose date, the first dose date will be used.
  - If the month and year are before the month and year of the first dose date, the last day of the month will be assigned to the missing day.
  - If the month and year are after the month and year of the first dose date, the first day of the month will be assigned to the missing day.
  - (2). Missing day and month
    - If the year is the same as the year of the first dose date, the first dose date will be used.
    - If the year is prior to the year of the first dose date, December 31 will be assigned to the missing fields.
    - If the year is after the year of the first dose date, January 1st will be assigned to the missing fields.
  - (3). Missing day, month, and year (or only year)
    - Do not impute.

#### Missing Data Imputation for Missing Concomitant Medication Stop Date

If the start date is non-missing and the imputed stop date is before the start date, the start date will be used. If the death date is available and the imputed stop date is after the death date, the death date will be used.

- (4) Missing day only
  - The last day of the month will be assigned as the missing day.
- (5) Missing day and month
  - December 31 will be assigned to the missing fields.
- (6) Missing day, month, and year
  - Do not impute.

#### 5.3.3. Missing/Partial Dates during Screening Visit

The following rules apply to dates recorded during the screening visits (e.g., prior therapies/medications, initial diagnosis):

- (1) Missing day only
  - The first day of the month will be used if the year and the month are the same as those for the first dose of study drug. Otherwise, the 15th will be used.
- (2) Missing day and month
  - If the year is the same as the year of the first dose of study drug, the 15th of January will be used unless it is later than the first dose, in which case the date of the first of January will be used.
  - If the year is not the same as the year of the first dose of study drug, the date of the first of July will be used, unless other data indicates that the date is earlier.
- (3) Missing day, month, and year
  - No imputation will be applied.

#### 5.3.4. Missing/Partial Dates in Post-study Anticancer Therapy

#### Post-study therapy/radiotherapy start date:

If the stop date is non-missing and the imputed start date is after the stop date, the stop date will be used as the start date.

- If year is missing (or completely missing), do not impute.
- If year is present and month and day are missing:
  - If year is the same as the year of last dose date, impute as the last dose date + 1.
  - If year is greater than the year of last dose date, impute as January 1<sup>st</sup>.

- If year and day are present and month is missing:
  - If year is the same as the year of last dose date, and day is not greater than the day of last dose date, impute the month as the month of last dose date + 1.
  - If year or day is greater than the year or day of last dose date, impute the month as the month of last dose date.
- If year and month are present and day is missing:
  - If year and month are the same as the year and month of last dose date, impute as last dose date + 1.
  - If year or month is greater than the year or month of last dose date, impute day as first day
    of the month.

#### Post-study therapy/radiotherapy end date:

If the start date is non-missing and the imputed stop date is before the start date, the start date will be used. If the death date is available and the imputed stop date is after the death date, the death date will be used.

- If year is missing (or completely missing), do not impute.
- If (year is present and month and day are missing) or (year and day are present andmonth is missing, impute as December 31st.
- If year and month are present and day is missing, impute day as last day of the month.
- If the imputed end date is earlier than the observed/imputed post-study therapy/radiotherapy start date, the end date will be imputed as the same as the start date.

#### 5.3.5. Missing/Partial Last Dose Date

Missing/incomplete last dose date from the treatment discontinuation page will be imputed as follows:

- (1) Missing day only
  - If the treatment discontinuation reason is death, the death date will be used.
  - Else if the last available dosing date from dosing data matches the partial last dose date from the treatment discontinuation page, the last available dosing date will be used.
  - Else the first day of the month will be used.

#### (2) Missing day and month

- If the treatment discontinuation reason is death, the death date will be used.
- Else if the last available dosing date from dosing data matches the partial last dose date from the treatment discontinuation page, the last available dosing date will be used.
- Else January 1<sup>st</sup> will be used.

- (3) Missing day, month and year
  - If the treatment discontinuation reason is death, the death date will be used.
  - Else the last available dosing date will be used.

The imputed last dose date will be compared to the available study discontinuation date and the data cut off date. Then the earliest date will be used.

#### 5.3.6. Relationship and Severity Imputation Rules for Adverse Events

Imputation will not be made for data listings and datasets. Missing severity and relationship will not be imputed. All treatment-emergent AEs are expected to have non-missing severity (to toxicity grade) and relationship at the time of database lock.

# 6. DISPOSITION, DEVIATIONS AND PATIENT CHARACTERISTIC DATA

An overall patient disposition summary will be presented for all subjects to show the number of unique patients who entered the study.

In addition, patient disposition will be presented by Module 1a or 1b and by dose/schedule with percentages based on the safety population. The following information will be presented for disposition:

- Included in each analysis population (DLT evaluation, safety, Efficacy and PK)
- Ongoing/discontinued study treatment at the data cut off
  - Including reasons for discontinuation of treatment as per the eCRF
- Ongoing/withdrawn/completion from study at the data cut off
  - Including reasons for study termination as per the eCRF

Disposition data will be listed for all patients and will include patient status, date of discontinuation from treatment, date of withdrawal from study and reason for treatment discontinuation and study withdrawal. In addition, the number and percentage of subjects by country and site will be summarized.

#### **6.1.** Protocol Deviations

There is no per protocol analysis population defined for this study, therefore patients will not be excluded from the data analysis and reporting based on deviations.

Any important deviations discovered during the trial either through the data collected on eCRFs or monitoring visits/reports will be listed and summarized (when the total number of important deviations <=10, only listing will be provided). Deviation data may be exported into the database via third party data such as an excel file used by study monitors to track deviations (e.g., deviations collected via the clinical study management system, CTMS).

The following deviations will be considered important deviations:

- Patients who entered the study but did not fulfil the entry criteria.
- Treatment deviations such as wrong treatment received or incorrect dose during the study. Note, treatment delays or changes due to AE management are not considered treatment deviations. A review of relevant data may be required to confirm all important deviations in this category.
- Patients who received a prohibited concomitant treatment, including prohibited anti-cancer treatments.

Following review of all reported deviations and associated data and prior to database lock, other important deviation categories may be added. Only important deviations will be summarized.

# 6.2. Demographic and Baseline Characteristics

Demographics will be summarized by Module 1a or 1b and dose schedule for the safety population. Baseline demographic will include age at informed consent, age group (<65 and ≥65 years), gender, race, ethnicity, height (cm), weight (kg), BMI (kg/m²). Baseline characteristics will include primary tumor type and ECOG status.

# **6.3.** Genotype and Mutation Status at Enrollment

The genes and mutation status of patients based on local test at enrollment will be listed and summarized.

A patient may test positive for more than one mutation/gene and so will be included under each mutation/gene category for the baseline summary.

#### 6.4. Disease Characteristics

The following disease characteristics will be summarized based on the Safety Population:

#### Disease History:

- Time since initial diagnosis (in years)
- Time since presentation of metastatic disease
- Primary tumor type
- Histology and grade of disease at diagnosis
- Molecular pathology at baseline (biomarkers per NCCN guidelines or as determined by NGS, IHC, and/or FISH)

#### Prior Anti-Cancer Therapy:

- Number of prior lines of treatment
- Prior gemcitabine use
- Prior use of platinum containing regimen
- Information on last prior anticancer therapy:
  - Reason for administration (adjuvant, neoadjuvant, advanced/metastatic, etc)
  - Best response
  - Disease progression (yes, no)
  - Time since end of last treatment in months
  - Duration of last treatment
  - Reason for end of regimen

# 6.5. Medical History

Medical history will be coded using the latest version of Medical Dictionary for Regulatory Activities (MedDRA) and will be summarized for the Safety Population, using System OrganClass (SOC) and preferred term (PT). The table will include the number and percentage of subjects and will be sorted in alphabetical order by SOC and PT. A subject will only be counted once within a class. A listing of medical and surgical history will also be provided. In particular, cancer related medical history will be summarized by SOC and PT.

#### 6.6. Prior and Concomitant Medications

Prior and concomitant medications will be coded using the World Health Organization (WHO) Drug Dictionary. The number and percentage of patients will be tabulated by WHO drug generic term for the Safety Population.

All prior and concomitant procedures (including transfusions) will be recorded from the Screening through to the EOT visit.

Prior medications will include medications which started prior to the date of first dose of study treatment. A summary table will present the numbers and percentages of patients who received prior therapy, including prior systemic anticancer therapy, prior radiation, prior surgery, and best response to the prior therapy, if known. Concomitant medications will include medications which started or were ongoing at the date of first dose of study treatment through to 30 days after the last dose of study treatment, or to the start of subsequent anticancer therapy, whichever occurs first. For Concomitant medications (including transfusions), the generic name of the drug (or trade name for combination drugs) must be specified along with the reason for use, and duration of treatment.

Details of prohibited concomitant medications are provided in the protocol. To determine prohibited medications programmatically, a coded list of all prohibited medications will be available prior to database lock. Listings of prior and concomitant medications will display a flag for prohibited medications. This information will be used to identify protocol deviations.

#### 7. SAFETY AND EXPOSURE DATA

Safety and tolerability will be assessed in terms of AEs, TEAEs, SAEs, DLTs, concomitant medications, PEs, vital sign measurements, clinical safety laboratory evaluations (hematology, serum chemistry, and urinalysis), ECOG performance scores, and ECGs including QTc.

Toxicity will be assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 unless otherwise specified. A toxicity will be considered dose-limiting if it occurs during the first 21 days, it is deemed to be related to treatment and it meets the criteria defined in Appendix 1. The **DLT Evaluable Population** will be used as the analysis set during dose escalation to make dose decisions in determining the MTD/RP2D. By-subject listings will be provided for DLTs (Cycle 1) using **DLT Evaluable Population**.

DLTs will be identified from the AE eCRF where the AE is selected as a DLT. All AEs reported as DLTs on the eCRF will be included even if they were not considered DLTs by the Safety Review Committee (SRC) during the study reviews. A listing of AEs considered DLTs by the SRC will be documented through SRC reports.

The MTD for this study will be defined as the highest dose with the toxicity probability (DLT rate) <25%. The BOIN drug combination design will be employed to find the MTD of continuous RP-6306 (Module 1a) or intermittent RP-6306 (Module 1b) in combination with gemcitabine. Each module will be evaluated separately. The target toxicity rate is 25%. Simulations confirm that with this study design, defining the MTD this way is equivalent tousing an isotonic regression with a descending pooled adjacent violators algorithm, which is the recommended method in the publication for BOIN study designs (Yuan et al., 2016).

#### 7.1. Adverse Events

Adverse events (AEs) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 24.0 or more recent version (at the time of database lock) and graded according to NCI-CTCAE version 5. All laboratory test results will be classified for toxicity grade according to the NCI-CTCAE version 5 criteria.

DLTs will be listed and summarized based on the DLT Evaluable Population.

Treatment emergent adverse events (TEAEs) are those events that occur or worsen on or after the first dose of study drug up through 30 days post the last dose. Those events occurred after start of subsequent anticancer therapy will be excluded.

An overview summary table of the number and percentage of patients in each of the categories listed below will be presented. This summary will be presented based on all patients in the study (overall summary to summarize unique patients) and then repeated split by module 1a or 1b and dose/schedule (see Section 5.1 for general presentation format).

- All TEAEs
- Treatment related TEAEs (related to either study drug)
- DLTs
- TEAEs with ≥ CTCAE Grade 3

- Treatment-related TEAEs with ≥ CTCAE Grade 3 (related to either study drug)
- Serious TEAEs
- Treatment-related serious TEAEs (related to either study drug)
- TEAEs with outcome of death
- TEAEs leading to discontinuation of study treatment
- TEAEs leading to dose reduction, dose interruption of study treatment

TEAEs will be summarized by system organ class (SOC), preferred term (PT), and by NCI CTCAE toxicity grade (where applicable). For summary tables, an AE that occurs more than once within a SOC and/or PT for the same patient will be counted only once using the worst NCI toxicity grade experienced.

Number and percentage of participants with TEAEs will also be presented by PT only. This summary will be sorted in decreasing order of frequency based on overall safety population.

For the summary tables related to toxicity grades, if there are two or more TEAEs (or AEs) with same SOC or PT and different toxicity CTCAE grades for the same subject, only the maximum toxicity grade of AE be counted.

Data listing will be provided for all TEAEs, TEAEs with ≥ CTCAE Grade 3 and serious TEAEs.

An AE table of most frequently occurring TEAEs, showing all events in at least 5% of patients, will be summarized by preferred term, by decreasing frequency based on all patients. This cut-off may be modified after review of the data.

TEAEs with outcome of death, leading to discontinuation of study treatment or leading to dose reduction, dose interruption or discontinuation of study treatment will be summarized by preferred term. Corresponding listings will be provided. If the number of occurrences is low (e.g., when  $\leq$  5 patients involved), only listing will be provided. If necessary, tabulated by preferred term depending on the number of TEAEs reported for those categories.

For patients who have a dose modification, all AEs (due to drug or otherwise) will be assigned to the initial dose group for summarizing. Any AE occurring before the first dose of study treatment will be included in the data listings but will not be included in the summary tables of AEs.

Summary tables will include only treatment-emergent adverse events (TEAEs). Non-TEAEs will be listed but will not be included in the summaries. Note that those events with onset after start of subsequent anticancer therapy will be excluded from the TEAE summary.

In addition, all treatment related SAEs will be summarized including all related SAEs with onset after the study treatment initiation, without using the TEAE window. Those events occurred after start of subsequent anticancer therapy will be excluded. The related SAEs will be summarized by PT. A listing of those related SAEs beyond the TEAE window will be presented.

A listing of all deaths and causes of deaths will be provided.

# 7.2. Treatment Exposure

Exposure will be derived for RP-6306 and gemcitabine respectively.

Duration of Exposure for each drug will be defined as the duration between the first and last doses of respective study drug

- Duration of RP-6306 exposure = last dose date first dose date + 1.
- Duration of gemcitabine exposure = last infusion date first infusion date + 7.

The last dose date will be obtained from the end of treatment (EOT) CRF page for each study drug.

Total duration of treatment for the study regimen is defined as Date of Treatment Discontinuation (from EOT page in the CRF) – first dose date +1. If treatment is still ongoing, use cut off date. If Date of Treatment Discontinuation is not collected, use the duration of exposure calculated above (take the longer of either drug).

Total dose received (mg) is the sum of total doses (mg) received. If a patient had a dose reduction/change during treatment, then the total dose received will be calculated for each actual dose received and then summed to give the total dose received.

Total dose received:  $\sum_{i=0}^{k}$  number of days dosed at dose  $x_i * dose x_i$ 

for i = 1 to k where i represents the number of dose levels received and k = number of distinct dose levels

Total planned dose will be derived as initial assigned dose a patient will receive without any interruptions or reductions based on the time-period between the date of first dose and date of last dose after excluding days when dosing information is not available, accounting for the number of treatment days per week. This is assuming the days without dosing information is missing at random.

Dose intensity will be derived as:

Dose intensity = (total dose received/total planned dose)\*100%

A dose interruption will be defined as a planned interruption where a decision is made to interrupt the dose temporarily, usually due to AE reason. Dose interruptions will be captured on the eCRF.

A dose reduction is any reduction prescribed by PI in dose/schedule compared to the initial dose.

Patients who do not have an end of treatment date in the eCRF at the time of analysis and reporting will be considered ongoing treatment. For deriving exposure, ongoing patients will be assumed to be ongoing at the date of the data cut off and therefore the data cut off date will be used to derive exposure.

Exposure will be listed and summarized by the Safety Population and presented by module 1a and 1b and dose/schedule.

The following will be presented

- Duration of exposure for each drug and overall
- Number and % of patients with at least 1 cycle, with at least 2 cycles...etc.
- Number of cycles treated (completed)
- Total dose received (mg)

- Dose intensity of RP6306 based on initial planned dose (%)
- Number and % of patients with at least one dose interruption reported in dosing log by considering only those incidences when AE is indicated as a reason
  - Further broken down by number with 1, 2 or  $\geq$  3 interruptions
  - Number and % of patients with dose interruption in Cycle 1, 2 or  $\geq$  3
- Number and % of patients with at least one dose reduction reported in dosing log considering only those incidences when AE is indicated as a reason
  - Further broken down by number with 1, 2 or  $\geq$  3 reductions
  - Number and % of patients with dose reduction in Cycle 1, 2 or  $\geq$ 3
- Number of patients with any dose escalation per protocol

Patients with both an interruption and reduction will be included in both the interruption and reduction summaries.

# 7.3. Laboratory Evaluations

All laboratory data recorded in the eCRF will be listed. Out-of-reference range values will be flagged as high (H) or low (L) in the listings. The results in conventional unit will be used in the summary tables.

Box plots for mean changes from baseline over time for selected lab parameters (hemoglobin, neutrophils, white blood cells [WBC], platelets, ALT, AST, BUN, total bilirubin, and creatinine) will be produced by module 1a or 1b and dose/schedule based on the safety population and the number of patients with data at the relevant timepoints. Sample size for each timepoint will be displayed.

Summary tables of actual and change from baseline from all the numerical lab tests will be provided.

Selected laboratory assessments (hemoglobin, neutrophils, white blood cells [WBC], platelets, ALT, AST, BUN, total bilirubin, and creatinine) will be also presented in shift tables showing baseline grade vs. maximum grade on study for lab assessment with CTCAE grading, based on all post-baseline data including unscheduled assessments. The denominator for each on-treatment maximum grade is the total number of patients in the corresponding row for baseline grade (i.e., the baseline row totals). The shift from baseline to worst value will be summarized.

For lab assessments which do not have CTCAE grading these will be categorized as low/normal/high based on reference ranges and shift tables will present baseline versus worst value on study.

If worst criteria could be a low or a high value or an increase or decrease (i.e., in both directions) then shift tables should be split to show shift from baseline to worst low/decrease value and then repeated for worst high/increase value. For example, CTCAE grade criteria is given for both lymphocytes count increased and lymphocyte count decreased.

Table 3: Clinical Safety Laboratory Analytes Collected in the Study

| Hematology | Serum Chemistry | Urinalysis |
|---|---|---|
| white blood cell count with differential (including at minimum: neutrophils, basophils, eosinophils, lymphocytes, monocytes) red blood cell count hemoglobin hematocrit platelet count | albumin alkaline phosphatase ALT AST BUN or urea calcium chloride creatinine glucose lactate dehydrogenase phosphate potassium sodium magnesium total bilirubin direct bilirubin total protein uric acid | specific gravity leukocyte esterase ketones protein glucose nitrite occult blood microscopy (if clinically indicated) pH |

Abbreviations: ALT = alanine aminotransferase; AST = aspartate aminotransferase; BUN = blood urea nitrogen

Post-baseline liver function tests including unscheduled assessments will be summarized in the following categories in Safety Population. A listing maybe used instead of summary table when the number of cases are few (<=5 patients)

- AST  $> 3 \times ULN$  or  $3 \times Baseline$  (if baseline value is >ULN)
- ALT  $> 3 \times ULN$  or  $3 \times Baseline$  (if baseline value is >ULN)
- ALP  $> 3 \times ULN$  or  $3 \times Baseline$  (if baseline value is >ULN)
- Total bilirubin > 2 × ULN

# 7.4. Vital Signs and Abnormalities

Descriptive statistics of pulse/heart rate, blood pressure (systolic and diastolic) (sitting/semi-recumbent), weight, and body temperature values will be summarized at baseline and post baseline visits, and changes from baseline will be summarized for post baseline visits based on the Safety Population. A separate listing will include all the vital sign measurements, including those from the unscheduled visits.

The following post-baseline vital signs will be summarized based on the Safety Population:

- Maximum post-baseline in SBP:
  - No increase

- Increase < 20 mmHg</li>
- Increase  $\ge 20$  mmHg
  - ≥ 160 mmHg and increase ≥ 20 mmHg
- Maximum post-baseline in DBP:
  - No increase
  - Increase < 20 mmHg</li>
  - Increase  $\ge$  20 mmHg
    - ≥ 100 mmHg and increase ≥ 20 mmHg

For the number of subjects meeting each category for the post-baseline results or for the change from, the numerator is the number of subjects with meeting the criterion at any post-baseline including the unscheduled and the denominator is the number of subjects with normal baseline and at least one post baseline assessment including unscheduled visits in the Safety Population.

A listing for patients with any post-baseline potentially clinically significant changes listed above will be also presented.

Box plots for changes from baseline over time for weight, DBP and SBP will be produced based on all patients in the Safety Population to identify signals of interest and showing the number of patients with data at the relevant timepoints.

#### 7.5. 12-lead ECG

Descriptive statistics (n, mean, SD, median, minimum, and maximum) of ECG parameters, including PR interval, RR interval, QRS duration, QT interval, and QTcF interval (Fridericia's corrections) will be presented for baseline, eachpost-baseline visit, and change from baseline to each post baseline visit for Safety Population. All measurements, including those during unscheduled visits, will be provided in data listings, but only the scheduled measurements will be included in the by-visit summary. The average of triplicate 12-lead ECG results will be used for descriptive statistics.

Overall ECG interpretation category (normal, abnormal NCS (not clinically significant), abnormal CS (clinically significant), and not evaluable) is collected in the CRF at baseline and each scheduled post-baseline visit. Shifts in ECG interpretation at baseline to worst post baseline as well as last value during the treatment period (up to last dose date for last value) will be presented. For triplicate 12-lead ECG results collected at a visit, the average of triplicate 12-lead ECG results will be used as the interpretation at baseline as well as post-baseline.

The QTcF will be categorized into the following categories.

- QTc interval >450 msec and ≤480 msec
- QTc interval >480 msec and ≤500 msec
- QTc interval >500 msec
The change from baseline in QTcF will also be categorized separately as follows:

- QTc interval increases from baseline by >30 msec and ≤60 msec
- QTc interval increases from baseline by >60 msec

For the number of subjects meeting each category for the post-baseline results, the numerator is the number of subjects with meeting the criterion at any post-baseline including unscheduled visits and the denominator is the number of subjects with normal baseline and at least one post baseline assessment including unscheduled visits in the Safety Population. For the number of subjects meeting each category for the change at post-baseline from baseline, the numerator is the number of subjects with meeting the criterion at post-baseline and the denominator is the number of subjects with baseline and at least one post baseline assessment in the Safety Population.

Box plots for absolute and change from baseline for QTcF will be produced based on all patients in the Safety Population to identify signals, displaying the number of patients with data at the relevant timepoints. All ECG parameters will be listed in a data listing. All ECG tables and listings will be reported on the safety analysis set.

A separate analysis on correlation between exposure and QTc will be performed as part of the population PK/ER analysis (outside the scope of this SAP).

# 7.6. Physical Examination and ECOG Performance Status

Abnormalities identified from physical examination will be listed for the safety analysis set.

Shift table of baseline ECOG performance to worst post-baseline status will be summarized as the number and % of patients in each ECOG category based on the Safety Population.

Any change in PE findings assessed as clinically significant should be recorded as an AE or SAE.

#### 8. EFFICACY DATA

The efficacy analysis will be summarized by dose regimen. Data from the backfill cohorts will be pooled with patients from the Dose Finding Phase that were treated at the RP2D.

Efficacy data will be summarized using the Efficacy Population, the selected analysis will be summarized by modified efficacy population.

# 8.1. Derivation of Efficacy Endpoints

## 8.1.1. Best Percentage Change in Tumor Size

Best percentage change in tumor size is defined as the largest decrease or smallest increase (in the absence of a decrease) in the sum of diameters of the TLs prior to progression or last evaluable assessment in the absence of progression.

• If a patient receives another anti-cancer therapy prior to progression, then data up until the least evaluable TL assessment prior to the start of subsequent therapy will be included

• If a patient does not have any evaluable post-treatment TL assessments to allow a derivation of best percentage change from baseline, they will be excluded from analysis

#### 8.1.2. Objective Response Rate (ORR)

Objective Response Rate (ORR) is defined as the proportion of patients with a confirmed response of CR or PR (i.e., 2 visit responses of either CR or PR at least 4 weeks apart) according to RECIST v1.1 criteria. This analysis will be limited to patients with measurable disease.

• Response will be assessed based on all evaluable assessments up to and including progression per RECIST v1.1. Responses occurring following subsequent anti-cancer therapy will be excluded from the assessment of ORR but will be included in the listing.

#### 8.1.3. Best Overall Response Rate

Best Overall Response Rate is defined as the proportion of patients with confirmed or unconfirmed response of CR or PR based on best overall response by investigators across all visits. Unconfirmed CR or PR will be defined as those patients with CR or PR only reported once in overall tumor assessment form by the Investigators according to RECIST 1.1.

CA-125 response is defined as having  $\geq$ 50% reduction from baseline, confirmed at the next assessment of at least 4 weeks later. Only those patients with baseline CA-125 > 2 times upper limit of normal (reference range is 0-35 kU/L) will be considered evaluable for CA-125 response.

Note that the unconfirmed CR or PR (assessed by investigator) is added as a response criterion in addition to protocol defined confirmed CR or PR, to identify signal of anti-tumor activity for the treatment.

## 8.1.4. Clinical Benefit Rate (CBR)

CBR is defined as the proportion of patients with a best overall response of CR or PR according to RECIST v1.1 based on Investigator's assessment, or ovarian patients with tumor marker response (GCIG for CA-125), or duration on treatment of at least 16 weeks without evidence of progression.

CRB will be defined for patients in efficacy populations.

#### 8.1.5. Tumor marker response

Tumor marker response (only for ovarian with abnormal baseline CA-125) is defined as having  $\geq 50\%$  reduction from baseline in CA-125 and confirmed in next assessment based on GCIG criteria.

#### 8.1.6. Duration of Response (DOR)

Duration of Response (DOR) will be derived for patients with a confirmed CR or PR only. DOR is defined as the time from the date of the earliest qualifying response (CR or PR) to the date of disease progression or death (if within 12 weeks after last adequate tumor assessment), whichever occurs earlier. Note, the end of response should coincide with the date of progression or death from any cause used for the PFS endpoint.

Given responses are required to be confirmed, the date of earliest qualifying response is the latest date for the visit where the initial overall visit assessment of CR/PR was observed rather than the confirmation visit assessment.

For patients who are alive or death beyond 12 weeks after last adequate tumor assessment without disease progression following response, DOR will be censored on the date of the last evaluable tumor assessment.

Table 4 gives the details rules of defining censoring/event for DOR.

Table 4: Censoring rule for Duration of Response (DOR) based on radiographical tumor assessment or death

| Situation | Date of Censoring or<br>Date of Event | DOR (weeks) | Censor |
|---|---|---|---|
| Documented disease progression (PD) before data cutoff date | Date of first PD | (Date of first PD – Date of first PR/CR + 1)/7 | 0 |
| No PD, but death date<br>before data cutoff date<br>and death date within 12<br>weeks after last adequate<br>tumor assessment | Date of death | (Date of death – Date of first PR/CR + 1)/7 | 0 |
| No PD and no death<br>before data cutoff date,<br>or death date beyond 12<br>weeks after last adequate<br>tumor assessment | Date of last adequate<br>tumor assessment <sup>a</sup> before<br>data cutoff | (Date of last adequate tumor assessment <sup>a</sup> – Date of first PR/CR + 1)/7 | 1 |

<sup>&</sup>lt;sup>a</sup> Adequate disease assessment is defined as a response assessment other than "not assessed" or "not evaluable."

## 8.1.7. Categorization of Best Tumor Response

For supportive information, the following confirmed best response categories will be derived for all patients with at least one post-baseline tumor assessment:

- Complete Response (CR): 2 visit responses of CR at least 4 weeks apart.
- Partial Response (PR): 2 visit responses of PR at least 4 weeks apart.
- Stable Disease (SD): If not confirmed CR/PR, at least one visit response of SD (or better i.e., unconfirmed CR/PR) recorded at least 6 weeks after the date of first dose of study drug.
  - To allow for the protocol window of  $\pm$  7 days, an overall assessment of SD on or after day 35 (i.e., 5 weeks) will be regarded as stable disease.
- Progressive Disease (PD): If not CR/PR/SD, and with at least one response of disease progression
- Not-Evaluable (NE): No evidence of CR, PR, SD, or PD. Either by default or the only visit response recorded is 'NE'.

## 8.1.8. Change in Tumor Size

The percent change in target lesions (TL) size compared to baseline will be derived at each visit as:

• Percent change in TL at Visit X = [(Visit X TL sum of diameters – Baseline TL sum of diameters)/Baseline TL sum of diameters] \*100

The best percent change will be derived as the largest decrease or smallest increase (in the absence of a decrease) up to and including progression or last evaluable assessment in the absence of progression. If a patient receives another anti-cancer therapy prior to progression, then data up until the last evaluable TL assessment prior to the start of subsequent therapy will be included.

Note that only TLs matched with baseline will be used for calculation of percent change.

## 8.1.9. Progression Free Survival (PFS)

Progression-Free Survival (PFS) is defined as the time from the first day of study drug administration (Day 1) to disease progression as defined by RECIST v1.1 criteria or death from any cause.

TL, NTL and new lesion assessments may be performed on different dates. The following rules will be applied for determine progression and censoring dates:

Date of progression will be determined based on the earliest of the dates of the component that triggered the progression. For example, if progression was due to a new lesion only then the date of the new lesions would be used. If progression was due to TLs and a new lesion, then the earliest of the TL and new lesion dates would be used.

Patients who are alive and free from disease progression will be censored at the date of their last evaluable tumor assessment prior to or equal to the data cut off date.

Any patient who dies in the absence of progression after 2 or more missed assessments will be censored at the date of their last radiographic tumor assessment. Specifically, if the death date is >12 weeks from the last tumor assessment, the death date will not be used for the calculation of PFS.

If a patient has no baseline tumor assessment/no post dose tumor assessments then they will be censored at 0 days for PFS, unless they died within 12 weeks from the date of first dose (and also before cut-off), in which case their death date will be used as a PFS event.

Table 5 gives the details rules of defining censoring/event for PFS.

PFS at 6 months will be reported based on KM methods as the number and % of patients estimated to be progression free at 6 months.

Table 5: Censoring Rule for time-to-event analyses (PFS) based on radiographical tumor assessment or death

| Situation | Date of Censoring or Date of<br>Event | Censor |
|---|---|---|
| Documented disease progression (PD) before data cutoff | Date of first PD | 0 |
| No PD, but death date is within 12 weeks from the last adequate post-baseline assessment <sup>a</sup> | Date of death | 0 |
| No PD, no post-baseline assessment, and death date is within 12 weeks from the date of first dose | Date of death | 0 |
| No PD, no post-baseline assessment <sup>a</sup> , and death date > 12 weeks from the date of first dose | Date of the first dose | 1 |

| Situation | Date of Censoring or Date of<br>Event | Censor |
|---|---|---|
| No PD, no post-baseline assessment <sup>a</sup> , and no death | Date of the first dose | 1 |
| No PD, Death date > 12 weeks from the last adequate post-baseline assessment <sup>a</sup> (e.g., 2 or more consecutive missed scheduled disease status assessments and the gap > 12 weeks) | Date of last adequate tumor assessment <sup>a</sup> | 1 |
| No PD or death, but with last adequate assessment <sup>a</sup> before data cut off | Date of last adequate tumor assessment <sup>a</sup> | 1 |

<sup>&</sup>lt;sup>a</sup> Adequate disease assessment is defined as a response assessment other than "not assessed" or "not evaluable."

This Censoring Rule is used for the data after implementation of data cut off.

# 8.2. Efficacy Analysis Methods

For overall response rate, ORR, and CBR, the number and percentage of patients along with an exact binomial 95% confidence interval (CI), using the Clopper-Pearson method, will be presented.

Unless otherwise specified, summary of all efficacy endpoints will be provided separately for Module 1a and 1b patients based on initial dose level.

The assessment of tumor efficacy will be based on the measurements recorded by the investigator.

A summary of the best objective response will be presented which will include the number and percentage of patients with a best response of CR, PR, SD, PD and NE.

Time-to-event endpoints (DOR, PFS) will be analyzed using the KM method and results will be summarized by the 25th, 50th and 75th percentiles, if estimable, with associated 2-sided 95% CIs. KM plots will be provided. For PFS, the number (%) of patients with an event and the number (%) of patients censored will also be presented. The rate of PFS at 4 and 6 months will be derived from the corresponding Kaplan-Meier curves. The KM analyses for DOR may be replaced by descriptive summary of median, and quartiles with individual listing for responders if total confirmed responders are few and less than 10 patients.

Maximum reduction in tumor size will be summarized by n, mean, standard deviation, median, 25<sup>th</sup> quartile and 75<sup>th</sup> quartile, minimum and maximum. The spider plots displaying change in tumor size over time for each patient will also be provided for each module and dose/schedule group as described above.

In addition, waterfall plots showing the best percentage change from baseline (largest decrease or smallest increase in the absence of a decrease) in the sum of the TL sizes will be produced for each module by dose/schedule group indicating each patient' best objective response.

Swimmer plots will be produced for each module and dose/schedule group to show the duration of study treatment per patient with indicators for timing of response, progression or death, where applicable. Include information on tumor type and genotype for each patient.



Data listings will be provided for all patients with information on best response, CBR, DOR, and PFS status. Also, the listings for the percent change / best percent change form baseline in the sum of the TL sizes will also be presented.







# 11. INTERIM ANALYSIS

No interim analysis is planned for this study.

# 12. REFERENCES

Eisenhauer EA, Therasse P, Bogaerts J, Schwart LH, Ford R, Dancey J, Arbuck S, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer. 2009; 45(2):228-47.

Liu S, Yuan Y. Bayesian optimal interval designs for phase I clinical trials. Appl Statist. 2015;64(3):507-523.

Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016;22(17):4291-301

# APPENDIX 1. DEFINITION OF DOSE LIMITING TOXICITY (DLT)

DLTs are defined as follows:

## Treatment-Related Hematologic TEAEs:

- Grade 4 neutropenia lasting at least 7 days or Grade 4 neutropenia lasting < 7 days requiring the use of G-CSF
- Febrile neutropenia (defined as absolute neutrophil count [ANC] <1000 cells/ $\mu$ L with a single temperature of 38.3°C [101°F] or a sustained temperature of 38°C [100.4°F] for >1 hour)
- Grade 4 thrombocytopenia or Grade 3 thrombocytopenia associated with Grade ≥2 bleeding
  Grade 4 anemia or Grade 3 anemia requiring red blood cell (RBC) transfusion per local hospital guidelines

## <u>Treatment-Related Non-Hematologic TEAEs:</u>

- Any Grade 3 treatment-related TEAE of >24-hour duration
- Any Grade 4 treatment-related TEAE of any duration

Any toxicity, regardless of the NCI CTCAE grade, resulting in discontinuation, Cycle 1 dose reduction or treatment with less than 75% of planned doses, will be reviewed by the SRC and will be considered a DLT if the SRC determines the toxicity cannot be attributed to the patient's underlying disease, other medical condition, or concomitant medications. Any death not clearly due to disease progression or extraneous causes are DLTs.

The following events will not be considered a DLT:

- Grade ≥3 non-hematologic laboratory abnormalities that are not considered clinically relevant in the opinion of the Investigator or respond to medical intervention
- Grade 3 fatigue with duration <7 days and resolved to Grade ≤2, unless it recurs within the first cycle and is considered drug-related by the Investigator
- Grade ≥3 nausea/vomiting/diarrhea that has not been treated with optimal supportive care
- The use of red blood cell transfusion for anemia Grade <3 or the use of G-CSF for Grade <4 neutropenia based on institutional practice guidelines.

# APPENDIX 2. GYNECOLOGICAL CANCER INTERGROUP DEFINITIONS FOR RESPONSE AND PROGRESSION IN PATIENTS WITH OVARIAN CANCER

For patients with ovarian cancer with elevated CA-125 levels, response evaluation will include cancer antigen 125 (CA-125) in addition to Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 criteria as per Gynecological Cancer Intergroup (GCIG) criteria (Rustin 2011).

## **Definition of Response by CA-125**

- A ≥50% reduction in CA-125 levels from a pretreatment sample. The response must be confirmed and maintained for at least 3 weeks (note that GCIG recommends maintenance for at least 28 days; Patients can be evaluated for a CA-125 response only if they have a pretreatment sample that is at least twice the upper limit of the reference range and within two weeks before starting treatment.
- Intervening samples and the confirmatory sample must be less than or equal to the previous sample (within an assay variability of 10%).
- The date when the CA-125 level is first reduced by 50% is the date of the CA-125 response.
- A CA-125 complete response can occur if CA-125 levels fall to within the reference range.

## **Definition of Progression by CA-125**

- For patients with elevated CA-125 pre-treatment that normalizes or for patients with CA-125 in the normal range at baseline: CA-125 at least 2 times the upper limit of the reference range on 2 occasions at least 1 week apart.
- For patients with elevated CA-125 pre-treatment which never normalizes: CA-125 at least 2 times the nadir value on 2 occasions at least 1 week apart.
- Progressive disease (PD) by objective change in tumor size should always take precedence over changes in CA-125 should it occur first. If measurable disease is reducing in size but the CA-125 suggests progression the patient should remain on treatment.
- CA-125 progression will be assigned the date of the first measurement that meets the above criteria.

Note: CA-125 progression in the absence of radiographic or other clinical evidence of progression will not be sufficient criteria for treatment discontinuation in this study.

Patients are not evaluable by CA-125 if they have received mouse antibodies (unless the assay used has been shown not to be influenced by human antimouse antibody) or if there has been medical and/or surgical interference with their peritoneum or pleura during the previous 28 days.

# **Evaluation of Best Overall Response by Combined CA-125 and RECIST 1.1 Criteria**

- If patients have a CA-125 response but have PD by RECIST within 28 days of the CA-125 response, they will be classified as PD.
- Patients whose best response by RECIST is stable disease (SD) but who have a CA-125 response will be classified as CA-125 responders

• For a patient to be classified as a complete responder according to RECIST, CA-125 levels must be within the normal range

#### For Patient with Measurable Disease

| Target<br>Lesion* | Nontarget† | New<br>Lesion | CA 125 | Overall Best<br>Response | |
|---|---|---|---|---|---|
| CR | CR | No | Normal | CR | Best RECIST 1.1 response for |
| CR | Non-CR Non-PD | No | Not PD | PR | CR and PR also requires it to |
| CR | CR | No | PR but not normal | PR | be confirmed and maintained |
| CR | NE | No | PR | PR | for at least 28 days if response |
| PR | Non-PD or NAE | No | Not PD | PR | is primary end point |
| NAE | Non-PD | No | PR | PR | |
| PD or Nev | v >28 days from CA 1 | 25 PR‡ | PR | PR | |
| SD§ | Non-PD | No | PR | PR | |
| SD§ | Non-PD or NAE | No | Not PR and not PD | SD | |
| PD or Nev | v ≤28 days From CA | 125 PR‡ | PR | PD | |
| PD | Any | Yes or No | Any | PD | |
| Any | PD | Yes or No | Any | PD | |
| Any | Any | Yes | Any | PD | |
| Any | Any | Yes or No | PD | PD | |

<sup>\*</sup>Target lesions include up to 5 measurable lesions (2 per organ) as defined by RECIST 1.1.

#### For Patients without Measurable Disease

| CA 125 | Nontarget Lesions* | New Lesions | Overall Serological Response | Best Response for This<br>Category Also Requires |
|---|---|---|---|---|
| Response and Normalized | CR | No | CR | Confirmed and maintained |
| Response | Non-PD | No | PR | for at least 28 days |
| Normalized but no response | Non-CR/Non-PD | No | SD | |
| Non-PR/non-PD | Non-PD | No | SD | |
| PD | Any | Yes or No | PD | |
| Any | PD† | Yes or No | PD | |
| Any | Any | Yes | PD | |

<sup>\*</sup>Nontarget lesions include ascites and peritoneal thickening, which are not measurable according to RECIST.

Reference: Rustin GJS, Vergote I, Elizabeth E, Pujade-Laurane E, Quinn M, Thigpen T, et al; Gynecological Cancer Intergroup. Definitions for response and progression in ovarian cancer clinical trials incorporating RECIST 1.1 and CA 125 agreed by the Gynecological Cancer Intergroup (GCIG). Int J Gynecol Cancer. 2011; 21(2):419-2

<sup>†</sup>Nontarget lesions include ascites and peritoneal thickening which are not measurable according to RECIST 1.1.

<sup>‡</sup>Patients who have a CA 125 response that occurs more than 28 days from PD according to RECIST 1.1 are considered a PR, according to best response, but PD if the RECIST 1.1 PD is within 28 days of CA 125 response.

<sup>§</sup>The protocol should specify the minimum time interval between 2 measurements for classification as stable disease.

NE, Not evaluated; NAE, not all evaluated.

<sup>†</sup>Unequivocal progression in nontarget lesions may be accepted as disease progression.

CR, Complete response; PD, progressive disease; PR, partial response; SD, stable disease.

# APPENDIX 3. RESPONSE EVALUATION CRITERIA IN SOLID TUMORS, VERSION 1.1

## **Evaluation of Target Lesions**

**Complete Response (CR):** Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.

**Partial Response (PR):** At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.

**Progressive Disease (PD):** At least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progressions).

**Stable Disease (SD):** Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.

### **Evaluation of Non-Target Lesions**

Complete Response (CR): Disappearance of all non-target lesions and normalization of tumor marker level. All lymph nodes must be non-pathological in size (<10 mm short axis).

Note: If tumor markers are initially above the upper normal limit, they must normalize for a patient to be considered in complete clinical response.

**Non-CR/Non-PD:** Persistence of one or more non-target lesion(s) and/or maintenance of tumor marker level above the normal limits.

**PD:** Appearance of one or more new lesions and/or unequivocal progression of existing non-target lesions. Unequivocal progression should not normally trump target lesion status. It must be representative of overall disease status change, not a single lesion increase.

Although a clear progression of "non-target" lesions only is exceptional, the opinion of the treating physician should prevail in such circumstances, and the progression status should be confirmed at a later time by the review panel (or principal investigator).

#### **Evaluation of Best Overall Response**

The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). The patient's best response assignment will depend on the achievement of both measurement and confirmation criteria.

## For Patients with Measurable Disease (i.e., Target Disease)

| Target Lesions | Non-Target Lesions | New Lesions | Overall<br>Response | Best Overall Response when<br>Confirmation is Required* |
|---|---|---|---|---|
| CR | CR | No | CR | >4 wks. Confirmation** |
| CR | Non-CR/Non-PD | No | PR | >4 wks. Confirmation** |
| CR | Not evaluated | No | PR | |
| PR | Non-CR/Non-PD/not evaluated | No | PR | |
| SD | Non-CR/Non-PD/not evaluated | No | SD | Documented at least once 8 wks. from first dose of study medication** |
| PD | Any | Yes or No | PD | No prior SD, PR or CR |
| Any | PD*** | Yes or No | PD | |
| Any | Any | Yes | PD | |

Abbreviations: CR = complete response; PD = progressive disease; PR = partial response; RECIST = Response Evaluation Criteria in Solid Tumors; SD = stable disease.

#### For Patients with Non-Measurable Disease (i.e., Non-Target Disease)

| Non-Target Lesions | New Lesions | Overall Response |
|--------------------|-------------|------------------|
| CR | No | CR |
| Non-CR/non-PD | No | Non-CR/non-PD* |
| Not all evaluated | No | not evaluated |
| Unequivocal PD | Yes or No | PD |
| Any | Yes | PD |

Abbreviations: CR = complete response; PD = progressive disease; SD = stable disease.

Reference: Eisenhauer EA, Therasse P, Bogaerts J, et al. New response evaluation criteria in solid tumors: revised RECIST guideline (version 1.1). Eur J Cancer 2009;45(2): 228–247.

<sup>\*</sup> See RECIST 1.1 manuscript for further details on what is evidence of a new lesion (Eisenhauer 2009).

<sup>\*\*</sup> Only for non-randomized trials with response as primary endpoint.

<sup>\*\*\*</sup> In exceptional circumstances, unequivocal progression in non-target lesions may be accepted as disease progression. Note: Patients with a global deterioration of health status requiring discontinuation of treatment without objective evidence of disease progression at that time should be reported as "symptomatic deterioration." Every effort should be made to document the objective progression even after discontinuation of treatment.

<sup>\*</sup>Non-CR/non-PD' is preferred over 'stable disease' for non-target disease since SD is increasingly used as an endpoint for assessment of efficacy in some trials so to assign this category when no lesions can be measured is not advised.